CLINICAL TRIAL: NCT03886077
Title: The Study of Hepatitis Eradication Receiving Protease Inhibitor Administration
Brief Title: Study of Hepatitis Eradication Receiving Protease Inhibitor Administration
Acronym: SHERPA
Status: Recruiting | Type: Observational
Sponsor: Sentara Norfolk General Hospital (Other)
Responsible Party: Principal Investigator, Gerry Cruz, Financial Analyst, Sentara Norfolk General Hospital
Other Study IDs: 2-26-2019 1.2
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Morality
MeSH Terms: conditions — Coronary Artery Disease | interventions — glecaprevir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hepatitis C Negative Donor Hearts: Hearts for transplantation that are not infected with Hepatitis C. (Negative NAT)
- Hepatitis C Infected Donor Hearts: Hearts for transplantation that are infected with Hepatitis C. (Positive NAT).
  Interventions: Drug: glecaprevir/pibrentasivir

INTERVENTIONS:
Drug: glecaprevir/pibrentasivir — 12 weeks of oral open label glecaprevir/pibrentasivir (Dose 3 tablets daily per package label).
  Groups: Hepatitis C Infected Donor Hearts

SUMMARY:
This is a prospective, non-blinded cohort study that will assess the safety, tolerability, and antiviral efficacy of glecaprevir/pibrentasivir therapy given post-discharge to HCV-negative recipients of HCV infected donors. Patients who meet entry criteria will be enrolled while on the transplant waitlist. At the time of transplant, some donors will be HCV positive / NAT positive and some will not be infected. Enrolled patients who receive an HCV negative donor will serve as contemporaneous controls. All study subjects who receive an HCV positive organ will be confirmed to have acquired HCV infection and genotype will be assessed prior to treatment with therapy.

DETAILED DESCRIPTION:
4. STUDY PROCEDURES 4.1 Subject Enrollment The patient is considered to be enrolled when they sign study consent. This may be months or years prior to the date of transplantation and therefore all study patients will be asked to affirm consent at the time of transplantation. There are 2 non-randomized study groups: Those patients who receive a non-HCV donor and those who receive a donor with HCV infection. Subjects will re-sign the consent on the line reserved for this purpose at the time of the transplant.

If the patient presented with a hepatitis C donor heart decides not to take that heart, they would remain in the study and when a suitable heart is found (infected or not), they would be followed post-transplant in the study.

4.2 Study Procedures Following transplantation with an HCV infectious donor, HCV viral load (RNA assay) will be measured at days 3,7 and 14 days post-transplant. The HCV viral load assay is a routine FDA cleared laboratory test which is one of the standard labs available at Sentara Norfolk General Hospital. It involves a blood sample of 5 cc which is then processed in the lab. Based on prior work, it is likely that all transplant recipients with infectious donors will seroconvert within this time frame. If these patients remain negative for HCV RNA, it will be rechecked every month for a total of 6 months. This routine testing is covered by insurance as this is the clinical standard for donors with elevated risk (Public Health Service increased risk).

Once a patient seroconverts to HCV positive, insurance authorization for treatment will be sought for treatment with glecaprevir/pibrentasivir. Based on input from Dr. Michael Ryan of Gastroenterology, insurance carriers are approving therapy given the noted efficacy, low comparative cost and the recent FDA approval of this drug in renal and liver transplant recipients. The study treatment is oral glecaprevir/pibrentasivir, 3 tablets daily with food, for a total of 12 weeks. The medication will be paid by the patient's insurance prescription coverage.

Serial measurements of HCV NAT (every month) will be conducted including through 24 weeks post-transplant. In addition, coronary angiography plus coronary intravascular ultrasound will be conducted at 6-12 weeks post-transplant and at one-year post transplant which will allow careful evaluation for cardiac allograft vasculopathy. Of note, it has been the policy of the Sentara Heart Transplant program for more than 5 years to perform baseline (early post-transplant) and annual coronary angiography and coronary intravascular ultrasound, and regardless of study participation, all patients will undergo this standard of care surveillance.

Post-transplant standard of care visits include frequent routine clinic labs (comprehensive metabolic panel, hepatic function panel, CMV viral load by PCR, creatinine kinase, complete blood count, B-type natriuretic peptide (BNP), tacrolimus or cyclosporine level if appropriate, sirolimus level if appropriate.

4.3 Post-Treatment Assessments Patients will have clinical standard of care visits to the transplant clinic, typically monthly in the first 6 months following transplantation. HCV NAT testing will be obtained at each visit for patients who received an infected donor, along with standard of care testing including cardiac biopsies, echocardiograms, chest-x-rays and other needed assessments. NAT testing is standard of care for recipients of increased infectious risk donors.

A visit will be mandatory at 12 weeks following the last dose of glecaprevir/pibrentasivir to draw HCV NAT testing.

Failure of HCV treatment If HCV RNA ≥ LLOQ at end of treatment (12 weeks of therapy) or viral relapse occurs in the Post-treatment follow-up, consultation with infectious disease and hepatology will be obtained. Testing for HCV drug resistance will be performed and patient will be treated as clinically indicated by the AHF team in consultation with specialists. Patients will be followed in regard to outcomes and achievement of SVR-12 until this occurs, or the patient dies or otherwise withdraws from the study.

4.4 End of Study Subjects are considered to have completed the study at 1 year post-transplant or the 1 year cardiac catheterization / IVUS is conducted, whichever is later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the inclusion criteria specified below in order to be eligible for participation in this study

  1. Willing and capable of providing written informed consent
  2. Age ≥18 years
  3. On UNOS list as a candidate for heart transplant

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria cannot be enrolled in this study.

  1. Individuals under 18 years of age
  2. History of advanced liver disease, including active hepatitis B or C, detectable hepatitis B surface Ag, hepatitis B DNA, HCV RNA, or cirrhosis
  3. Pregnant individuals
  4. HIV antibody positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 subjects listed for cardiac transplantation will be enrolled. Patients will be educated about this protocol prior to transplant, and informed consent obtained. Enrolled subjects who receive a transplant with a NAT positive HCV infected donor will undergo NAT testing and surveillance post-operatively. In addition, patients who are offered an HCV infectious organ will be "re-consented" at the time of transplantation admission.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response at 12 weeks following therapy. | 12 weeks following completion of study drug.
  12 weeks after the completion of drug that the patient no longer has Hepatitis C.

SECONDARY OUTCOMES:
Coronary allograft vasculopathy at 1 year post transplant. | 1 Year post heart transplant.
  Presence of coronary disease at 1 year post heart transplant.

CONTACTS AND LOCATIONS:
Overall Officials: David Baran, MD, Principal Investigator — Sentara Norfolk General Hospital
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No